CLINICAL TRIAL: NCT06537336
Title: Optimizing Pulmonary Health and Quality of Life in Breast Cancer Survivors: A Randomized Controlled Trial Combining Incentive Spirometry and Aerobic Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hermina Hospitals (Industry)
Collaborators: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Geraldi Christian Candra, Principal Investigator, Hermina Hospitals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LB.02.01/X.6.5/76/2023
Record Dates: First submitted 2024-08-01; First posted 2024-08-05 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
Keywords: Aerobic exercise; Breast cancer; Incentive spirometry; Lung function; Quality of life
MeSH Terms: conditions — Breast Neoplasms | interventions — Respiratory Function Tests

STUDY DESIGN:
Intervention Model Description: The patients in the treatment group underwent aerobic and volumetric incentive spirometry breathing exercises. The control group performed only aerobic exercise. The aerobic exercise program was conducted over 8 weeks using a stationary bicycle. Patients were initially selected based on the inclusion and exclusion criteria, and informed consent was obtained. Before and after the intervention, lung function tests using spirometry and QoL measurements were conducted using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaires-Core30 (EORTC-QLQ-C30).
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): The patients in the treatment group underwent aerobic and volumetric incentive spirometry breathing exercises
  Interventions: Device: QoL; Device: lung function
- control group (Active Comparator): The control group performed only aerobic exercise.
  Interventions: Device: QoL; Device: lung function

INTERVENTIONS:
Device: QoL — QoL measurements were conducted using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaires-Core30 (EORTC-QLQ-C30).
Device: lung function — lung function tests using spirometry

SUMMARY:
Breast cancer survivors frequently experience diminished lung function and decreased quality of life (QoL) following radiation therapy (RT). Additionally, incentive spirometry, which encourages prolonged deep breathing, could potentially amplify lung function and QoL when paired with aerobic exercises. This study investigated the combined effect of aerobic and breathing exercises using incentive spirometry on lung function and QoL in patients with breast cancer after RT.

DETAILED DESCRIPTION:
Study Design This experimental study employed a single-blind randomized controlled trial design with two groups. Consecutive sampling was conducted based on the order of arrival. Group allocation (control group with aerobic exercise or treatment group with incentive spirometry breathing exercises combined with aerobic exercise) was determined using a simple random sampling method with a lottery. The data were analyzed using SPSS version 25.0.

Participants Participants were patients with breast cancer who had completed Radiotherapy at Hasan Sadikin General Hospital Bandung between April 2023 and June 2023.

Research Procedure Patients were initially selected based on the inclusion and exclusion criteria, and informed consent was obtained. Before and after the intervention, lung function tests using spirometry and QoL measurements were conducted using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaires-Core30 (EORTC-QLQ-C30). The EORTC-QLQ-C30 was designed to assess seven domains of QoL in cancer patients: physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning, overall health status, and symptom domains. The EORTC-QLQ-C30 questionnaire has been translated into Indonesian from Dyah A.P's research. and has shown validity scores >0.70 and reliability scores >0.80 in evaluating the QoL of cancer patients undergoing therapy.14 The patients in the treatment group underwent aerobic and volumetric incentive spirometry breathing exercises. The control group performed only aerobic exercise.

The aerobic exercise program was conducted over 8 weeks using a stationary bicycle. The training frequency was three times per week. Each session lasted 40 min, consisting of 5 min of warm-up, 30 min of main exercise, and 5 min of cool-down. The exercise intensity was moderate (RPE 12-13).

Volumetric incentive spirometry exercises were performed 15 min after completing the aerobic exercise. This exercise used sustained maximal incentive spirometry (Voldyne 5000®). The program was conducted over eight weeks with a training frequency of three times per week. Each session included five sets of exercises, with each set consisting of 10 breathing repetitions and a 1-minute rest between sets. The intensity of this exercise involved performing maximal inspiration from the residual volume (RV) to the total lung capacity (TLC) that the subject could achieve. The inspiratory volume reached was used as the target for subsequent training sessions.

ELIGIBILITY:
Inclusion Criteria:

* age between 30 and 59 years;
* diagnosis of histological breast cancer (AJCC Stage I to III) and completion of RT for > 3 months;
* hemoglobin level > 10 mg/dL;
* ability to comprehend verbal and written instructions;
* cooperative participants, willingness to participate in the study, and ability to engage in exercises by signing an informed consent form; and
* Nonreactive COVID-19 antigen swab test results.

Exclusion Criteria:

* cancer metastasis to the bone, lungs, or surrounding organs;
* aerobic exercise and incentive spirometry breathing exercises within the last six months;
* uncontrolled hypertension (blood pressure >140/90 mmHg on antihypertensive treatment);
* unstable cardiovascular diseases (including unstable angina, acute myocardial infarction, arrhythmias, severe valvular heart disease, severe arteriovenous stenosis, and decompensated congestive heart failure) determined from medical records, history, physical examination, and electrocardiograms;
* uncontrolled blood sugar level (random blood sugar >200 mg/dL or fasting blood sugar >126 mg/dL);
* acute or chronic respiratory diseases (asthma, chronic obstructive pulmonary disease, and pulmonary tuberculosis);
* neuromuscular dysfunction (spinal muscular atrophy, Guillain-Barré syndrome, and multiple sclerosis);
* degenerative arthritis;
* physical limitations affecting stationary cycling; and
* musculoskeletal disorders.

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — age between 30 and 59 years
Enrollment: 38 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
lung function | 8 weeks of exercises
  Lung function tests will be assessed using a spirometry. It measures the value of predicted forced vital capacity (FVC) and forced expiratory volume in one second/forced vital capacity (FEV1/FVC ratio). lower scores are associated with poor lung function
quality of life as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaires-Core30 (EORTC-QLQ-C30). | 8 weeks of exercises
  The EORTC-QLQ-C30 was designed to assess seven domains of quality of life in cancer patients: physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning, overall health status, and symptom domains. scores range from 0 to 100, with higher scores indicating better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Dian M Sari, dr, Study Chair — Padjajaran University
Locations (1):
- Padjajaran University, Bandung, West Java, Indonesia